CLINICAL TRIAL: NCT00561990
Title: A RANDOMIZED, MULTICENTER, PHASE IIB/IIIA STUDY OF GEMCITABINE AND THE MONOCLONAL ANTIBODY NIMOTUZUMAB (OSAG 101) VERSUS GEMCITABINE AND PLACEBO FOR THE TREATMENT OF CHEMOTHERAPY-NAIVE PATIENTS WITH LOCALLY ADVANCED OR METASTATIC PANCREATIC CANCER
Brief Title: Nimotuzumab in Adults With Pancreatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oncoscience AG (Industry)
Collaborators: Marienhospital Herne (Other); University of Kiel (Other); Gemeinschaftspraxis für Hämatologie und Onkologie, Köln, Germany (Unknown); Onkologisches Zentrum III, Medizinische Klinik, Mannheim, Germany (Unknown); Onkologische Gemeinschaftspraxis, Mülheim, Germany (Unknown); II. Medizinische Klinik u. Poliklinik, Klinikum rechts der Isar, München, Germany (Unknown); Hämatologisch-Onkologische Schwerpunktpraxis, Münster, Germany (Unknown); Praxis für Internistische Onkologie und Hämatologie, Recklinghausen, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: OSAG101-PCS07
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer, Advanced or Metastatic
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab (Active Comparator): Nimotuzumab
  Interventions: Drug: Nimotuzumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab

SUMMARY:
CHEMOTHERAPY-NAIVE PATIENTS WITH LOCALLY ADVANCED OR METASTATIC PANCREATIC CANCER

DETAILED DESCRIPTION:
Pancreatic cancer is responsible for 227.000 deaths per year, and is the eighth most common cause of death from cancer in both sexes combined, a position relatively high when compared to incidence (thirteenth position) because of the very poor prognosis (the M/I ratio is 98%) (Global Cancer Statistics, 2002). The incidence of pancreatic carcinoma has increased almost 300% since 1950 and now exceeds the incidence of stomach cancer and cancer of the rectum. Carcinoma of the exocrine pancreas is nearly always a fatal disease. The overall 5-year survival rate for the disease is 4.1%.

Locally advanced or metastatic pancreatic cancer is relatively unresponsive to chemotherapy. Gemcitabine therapy provides some benefit and modestly improves survival compared with fluorouracil, but median survival in patients with advanced disease remains less than 6 months (Burris et al, 1997). Cytotoxic drug combinations were not able to show survival advantage compared to Gemcitabine alone in numerous randomized phase III studies.

Altered expression or constitutive activation of the epidermal growth factor receptor (EGFR/HER1/erbB1) commonly occurs in both primary and metastatic pancreatic cancers and is often a critical factor in progressive growth and resistance to normal mechanisms of cell death. Epidermal growth factor receptor expression in pancreatic cancer has been correlated with tumor aggressiveness.

Clinical trials already suggest that EGF-R targeted therapy may improve the antitumor activity of chemotherapy for treatment of pancreatic carcinoma. Monoclonal antibodies specific to EGF-R can be combined safely and effectively with chemotherapy.

Nimotuzumab (OSAG101, hR3, Theraloc) is a humanized monoclonal antibody (mAb) that binds to the EGFR. In preclinical studies the antibody has shown potent antitumor activity. Based on phase I data, the recommended dose has been established at 200 mg weekly. A previous phase II study in children with high grade brain tumors showed activity of Nimotuzumab as a monotherapeutic agent, even in prognostic very unfavourable diffuse, intrinsic pontine glioma. No drug related side effects were reported.

Nimotuzumab (OSAG101, Theraloc) in combination with radiotherapy for treatment of locally advanced squamous cell carcinomas of the head and neck resulted in high rates of antitumor response, and was accompanied by a favourable safety profile. Nimotuzumab (OSAG101, Theraloc) has a high hepatic uptake level.

This randomized, placebo-controlled Phase IIb/IIIa study analyzes the efficacy and safety of Nimotuzumab in combination with Gemcitabine for the treatment of chemotherapy-naive patients with advanced unresectable or metastatic pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. written informed consent.
2. histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the pancreas not amenable to curative radiotherapy or surgery.
3. measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (ie, target lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral computed tomography [CT] scan).
4. able to take medications orally.
5. at least18 years of age or older.
6. Karnofsky Performance Status (KPS) ≥ 70% (see Appendix A).
7. life expectancy of > 12 weeks.
8. adequate organ function as defined by the following criteria:

   * Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal (ULN).
   * If liver function abnormalities are due to underlying liver metastasis, then AST (SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
   * Total serum bilirubin ≤ 3.0 times ULN (if due to underlying liver metastasis, then total bilirubin may be ≤ 5 times ULN).
   * Absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units (IU]).
   * Platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
   * Hemoglobin value ≥ 9.0 g/dL.
   * Calculated creatinine clearance ≥ 60 mL/min (based on serum creatinine) (Cockcroft Gault formula).
9. willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
10. both female and male patients must use adequate methods of contraception.

Exclusion Criteria:

1. had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Any prior anticancer chemotherapy.
   2. Radiation therapy to a target lesion unless there was evidence of PD after radiotherapy (and this target lesion must not be the only site of measurable disease).
   3. Any radiotherapy within the previous 3 weeks.
   4. Any investigational agent received either concurrently or within the last 30 days.
   5. Current enrollment in another clinical trial.
2. Major surgery within the previous 3 weeks.
3. Symptomatic brain metastasis not controlled by corticosteroids.
4. Leptomeningeal metastasis.
5. Previous or concurrent malignancy other than pancreatic cancer except adequately treated carcinoma in-situ of the cervix or non-melanoma skin cancer.
6. Uncontrolled ascites requiring drainage at least twice a week.
7. Other serious illness or medical condition(s) including, but not limited to, the following:

   * Uncontrolled congestive heart failure (New York Heart Association [NYHA]
   * Class III or IV, see Appendix F), angina pectoris, arrhythmias, or hypertension.
   * active infection.
   * known (at time of entry) gastrointestinal disorder, including malabsorption,
   * chronic nausea, vomiting, or diarrhea, present to the extent that it might interfere with oral intake and absorption of study medication.
   * Poorly controlled diabetes mellitus.
   * Psychiatric disorder that may interfere with consent and/or protocol compliance.
   * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
   * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
8. pregnant or lactating female.
9. known hypersensitivity to Anti-EGFR antibodies.
10. with reproductive potential who refuses to use an adequate means of contraception (including male patients).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression (TTP) and overall survival (OS) in chemotherapy-naive patients. To assess the efficacy of Nimotuzumab as add on therapy to Gemcitabine in comparison with Gemcitabine and placebo | Week 8, 12

SECONDARY OUTCOMES:
To evaluate the objective tumor response (overall response rate [ORR]) and duration of response (DR) To evaluate the safety profile of Nimotuzumab in combination with Gemcitabine To evaluate quality of life (QoL) according to EORTC | Week 8, 16

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Strumberg, MD, Principal Investigator — University Bochum
Locations (1):
- Marienhospital Herne, Herne, Germany

REFERENCES:
- [Derived] Schultheis B, Reuter D, Ebert MP, Siveke J, Kerkhoff A, Berdel WE, Hofheinz R, Behringer DM, Schmidt WE, Goker E, De Dosso S, Kneba M, Yalcin S, Overkamp F, Schlegel F, Dommach M, Rohrberg R, Steinmetz T, Bulitta M, Strumberg D. Gemcitabine combined with the monoclonal antibody nimotuzumab is an active first-line regimen in KRAS wildtype patients with locally advanced or metastatic pancreatic cancer: a multicenter, randomized phase IIb study. Ann Oncol. 2017 Oct 1;28(10):2429-2435. doi: 10.1093/annonc/mdx343. PMID 28961832